CLINICAL TRIAL: NCT01482780
Title: EASY-TRIAL: Evaluation of a Local Preconditioning Effect in Patients Undergoing Cardiac Surgery
Brief Title: Evaluation of a Local Preconditioning Effect in Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic reasons, lack of funding
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Mohl, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EASY-TRIAL
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Heart Disease; Coronary Artery Bypass Graft Triple Vessel
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICSO (Experimental): PICSO (pressure controlled intermittent coronary sinus occlusion), a special coronary sinus catheter will be introduced after induction of anaesthesia until going on bypass.
  Interventions: Device: PICSO
- Control (No Intervention): normal procedure of preparing Bypass grafts. Equivalent time before going on Bypass is determined as control period

INTERVENTIONS:
Device: PICSO — PICSO (pressure controlled intermittent coronary sinus occlusion) will be used in the pre ECC period. The procedure of PICSO will be performed in analogy to retrograde cardioplegia.
  Other Names: PICSO, Miracor medical Systems, Austria
  Arms: PICSO

SUMMARY:
The aim of the study is to analyze the potential of pressure controlled intermittent coronary sinus occlusion (PICSO) to prevent/reverse the ischemic burden as well as reperfusion injury. To achieve insight into the clinical significance of this local preconditioning effect, global hemodynamics, cardiac performance and clinical outcome in the first 30 days will be related to the ability of this intervention to protect the myocardium in elective surgical procedures, ameliorating cellular decay and preserving the microcirculation therefore improving graft flow, reducing enzyme leakage and finally improving myocardial performance.

DETAILED DESCRIPTION:
* Patients undergoing elective coronary artery bypass graft (CABG) will be enrolled in this study.
* A computerized randomization process is used to obtain similar distributions within each group. Stratification will be done by the severity of coronary artery disease, age and sex.
* Routine blood sampling will be performed the day before surgery as well as a transthoracic echocardiography (TTE) study to determine ventricular volumes and valvular function.
* A modified Minnesota quality of Life questionnaire will be assessed and these data will be compared with 30 days outcome data screened in an outpatient environment.
* A 12 lead electrocardiogram will be obtained. To assess eligibility and to assure grouping (stratification & randomization) patients will be scored using the additive EuroSCORE. Pre-, intra-, and postoperative (up to 72 hrs) measurements of myocardial enzyme leakage will be performed using standard diagnostic procedures (cardiac troponin T, CK-MB, and total creatine kinase), as well as serial electrocardiograms and echocardiograms.
* Perioperative infarction will be assessed as the development of new persistent regional wall motion abnormalities in echocardiography together with electrocardiographic alterations and CK-MB increases and new Q-wave PMI.
* Sequential cytokine analyses (IL-1, IL-6, IL-8, IL-10, IL-17, VEGF and TNF- alpha ) preoperatively, at the beginning of the operation, the beginning of ECC and 6,24 h and 30 days postop.
* Serial quantification of global and regional wall motion will be recorded using TEE measurements during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex and between 18 and 85 years of age scheduled for surgery without severe confounding disease will be asked to participate in the study.
* Written informed consent will be obtained in eligible patients.

Exclusion Criteria:

* Patients with unstable angina pectoris and/or myocardial infarction within the last 30 days, as well as persons with planned concomitant valvular interventions will be excluded. Patients with malignoma, severe hepatic, renal and pulmonary disease will also be excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Reduction in enzyme leakage measured by AUC. | 72 hours postop
  Enzyme leakage (Troponin T, CK-MB) will be measured preoperatively, at the beginning of the operation, the beginning of ECC at the time of reperfusion the arrival on the ICU and 6,12,24,48 and 72 hours postop and the area under the curve will be calculated (AUC until 72 hours).
  Study Hypotheses:
  1. PICSO reduces troponin T leakage about 30 % measured by AUC until 72h in comparison to controls.
  2. PICSO improves 30d and long-term outcome

SECONDARY OUTCOMES:
Combined endpoint of major adverse cardiovascular events (MACE) and mortality after 30 days. | 30 days
N-terminales pro brain natriuretic peptide (NT-pro BNP) values at 1 day pre-surgery as well as 30d and 6 months post-operative | 30 days
Pre-operative (1d) as well as post-operative (6, 12, 24, 48, 72 h, 30d) C-reactive protein (CRP) measurements | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Werner Mohl, DDr, Principal Investigator — Medical University of Vienna, Abteilung für Herz-, Thoraxchirurgie; Werner Mohl, DDr., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria